CLINICAL TRIAL: NCT04264299
Title: Comparative Study of Three Common Bile Duct Closure Techniques After Choledocholithotomy: Safety and Efficacy
Brief Title: Comparative Study of Three Common Bile Duct Closure Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Omar, Associate professor of HPB surgery, South Valley University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVU 300
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Common Bile Duct Closure
Keywords: choledocholithiasis; T-tube; primary repair; biliary stenting
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T tube drainage (Active Comparator): Closure of common bile duct after choledocholithotomy over T tube
  Interventions: Procedure: Primary closure; Procedure: Antegrade stenting
- Primary closure (Experimental): Primary closure of the common bile duct after choledocholithotomy
  Interventions: Procedure: T tube drainage; Procedure: Antegrade stenting
- Antegrade stenting (Experimental): Closure of common bile duct over antegrade biliary plastic stent
  Interventions: Procedure: T tube drainage; Procedure: Primary closure

INTERVENTIONS:
Procedure: T tube drainage — closure of common bile duct over T tube
  Arms: Antegrade stenting; Primary closure
Procedure: Primary closure — Primary closure of common bile duct
  Arms: Antegrade stenting; T tube drainage
Procedure: Antegrade stenting — Closure of common bile duct over antegrade plastic biliary stent
  Arms: Primary closure; T tube drainage

SUMMARY:
This study evaluates the efficacy and safety of three different methods of CBD repair after common bile duct exploration and provides more evidence for selecting the optimal duct closure after choledocholithotomy.

DETAILED DESCRIPTION:
At present, the commonest available options for CBD closure include repair over T-tube drain, primary closure, and repair after antegrade biliary stenting. All three methods present speciﬁc technical performance features, require different postoperative management protocols, and are charged with speciﬁc morbidity related to the procedure and therefore should not be considered the same procedure in the context of CBDE.

Repair over T-tube is the traditional surgical technique. It has many advantages as post-operative distal CBD decompression, trans-tubal cholangiography, and availability of retained CBD stones extraction. However, it has several potential complications up to 10% of patients. The most frequent complications are bile leakage, tract infection, T-tube dislodgement, electrolyte and nutritional disturbances, cholangitis, or acute renal failure from dehydration due to inadequate water ingestion. It also causes discomfort and persistent pain to the patient along with increased hospital admission and thus the economic burden to the country. Primary closure of CBD has been described in the literature to overcome these adverse consequences of the T-tube. However, it has many potential complications as a potential bile leak and CBD stricture, which may occur due to papillary edema and insufficient bile duct expansion. There are conflicting results regarding significant differences in the morbidity and mortality between primary closure and T-tube drainage. There is no conclusive evidence displaying whether primary closure is better or worse than T-tube drainage after CBD exploration.

Using a biliary stent in primary closure is an effective method to decrease the two complications, which can reduce biliary pressure without bile loss. Although there are some available drainage options after CBDE, a consensus on the optimal drainage is yet to be reached.

ELIGIBILITY:
Inclusion criteria

* CBD stones
* age from 20 to 80,
* CBD > 0.8 cm and < 2.5 cm,
* American Society of Anesthesiologists (ASA) grade I, II or III,
* agreement to randomization and complete the study requirement. Exclusion criteria
* acute suppurative cholangitis,
* acute biliary pancreatitis,
* biliary malignancy,
* biliary malformation,
* distal CBD stenosis and or obstruction,
* trans-cystic stone extraction,
* explorations followed by choledochojejunostomy and choledochoduodenostomy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Postoperative bile leak | 3rd to 7th postoperative day
  The discharge of fluid via intra-abdominal drain or intra-abdominal fluid with bilirubin concentration at least 3 times the serum bilirubin concentration measured at the same time on or after the 3rd postoperative day, or as the need for radiologic or surgical intervention because of biliary collections.
Post operative biliary stricture | 6 month
  The segmental shrunken of CBD diameter and proximal dilatation by MRCP.
Recurrent biliary stones | 6 month
  Common bile duct stone after 6 months of the procedure

SECONDARY OUTCOMES:
Visual analogue score | 3 days
  the severity of postoperative pain. from 0 (no pain) to 10 (maximum pain)
The number of patients need postoperative opioid | 3 days
  The patients need of postoperative opioid (pethidine Hcl 50 mg)
Postoperative bilirubin level | 7 days
  the rate of decreased bilirubin postoperatively
Hospital stays | 10 days
  the number of days in hospital from the day of operation to the day of discharge
Drain-carried time | 20 days
  the number of days before drain removal
Total cost of treatment | Through study completion, average 6 month
  The cost of intervention and management of postoperative complications
Return to normal activity | 30 days
  the number of days required for the patient to return to normal activity
Type of re-intervention | 6 month
  the number of intervention required for each patient totally

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A. Omar, Ass. Prof., Principal Investigator — South Valley University
Locations (1):
- Mohammed Ahmed Omar, Sohag, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omar MA, Redwan AA, Alansary MN. Comparative study of three common bile duct closure techniques after choledocholithotomy: safety and efficacy. Langenbecks Arch Surg. 2022 Aug;407(5):1805-1815. doi: 10.1007/s00423-022-02597-3. Epub 2022 Jul 4. PMID 35786738